CLINICAL TRIAL: NCT00897117
Title: Molecular Fingerprinting of Lung Cancer
Brief Title: Collecting and Analyzing Tissue Samples From Patients Undergoing Surgery for Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Grogan, Associate Professor of Thoracic Surgery, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC THO 0136; P50CA090949 (NIH); VU-VICC-THO-0136 (Other: VICC); P30CA068485 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gene Expression Profiling; Microarray Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Both prospective and retrospectives samples of blood and tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Resectable non-small cell lung cancer: Patients with clinical stage I or II invasive lung cancer that can be completely removed by surgery and who have not undergone chemotherapy or radiotherapy before surgery
  Interventions: Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: protein expression analysis; Other: biologic sample preservation procedure; Other: laboratory biomarker analysis; Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry

INTERVENTIONS:
Genetic: gene expression analysis — Blood and lung tissue collection
Genetic: microarray analysis — Blood and lung tissue collection
Genetic: protein expression analysis — Blood and lung tissue collection
Other: biologic sample preservation procedure — Blood and lung tissue collection
Other: laboratory biomarker analysis — Blood and lung tissue collection
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry — Blood and lung tissue collection

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that may occur in RNA and identify biomarkers related to cancer.

PURPOSE: This research study is collecting and analyzing lung tissue samples from patients undergoing surgery for non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop statistical and computational methods for modeling the relationships between multiple variable protein and RNA expression data and clinical endpoints using both supervised and unsupervised classification and pattern recognition approaches.
* Determine protein and RNA expression fingerprints on completely resected non-small cell lung cancer without prior chemotherapy.
* Correlate protein and RNA expression fingerprints with T-stage and nodal involvement at the time of surgery, and collect outcome data to allow correlation with recurrence (local and/or distant) and survival.

OUTLINE: This is a multicenter study.

Any excess tissues removed from surgery and would otherwise be discarded (tissues not used for diagnosis and/or treatment decision making) are obtained for this study. Tissue are analyzed for molecular features that predict biologic behavior. Quantitation of RNA, gene expression profiles, and protein expression patterns are assessed by matrix-assisted laser desorption/ionization time of flight mass spectroscopy and microarray analysis.

Medical records are reviewed to obtain information about results of tests associated with cancer diagnosis. Further progress in cancer treatment and tumor behavior after surgery are followed via record review.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of non-small cell lung cancer

  * Clinical stage I and II disease
  * Resectable disease and complete surgical resection planned
* Treated on companion studies at Vanderbilt University, the Veterans Administration hospital, St. Thomas, and Vanderbilt-Ingram Cancer Center Affiliate Network
* Tumor specimen samples must be available at resection

Exclusion criteria

* Chemotherapy before surgery
* Radiotherapy before surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have clinical stage I and II non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2001-05; Primary Completion 2031-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Protein and RNA expression fingerprints from collected samples | after collection of designated samples

SECONDARY OUTCOMES:
Development of statistical and computational methods to model relationship of data and clinical outcomes | after laboratory gene analysis work is completed
Correlation of protein and RNA expression fingerprints with recurrence (local and/or distant) and survival | after collection of designated samples

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grogan, MD, Principal Investigator — Vanderbilt Medical Center
Locations (3):
- United States (3):
  - Dan Rudy Cancer Center at Saint Thomas Hospital, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/